CLINICAL TRIAL: NCT01068990
Title: Detection and Characterization of Lower Respiratory Infections in Critically Ill Patients
Status: Recruiting | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sang-Ho Choi, Doctor, Asan Medical Center
Other Study IDs: AICUP
Record Dates: First submitted 2010-02-12; First posted 2010-02-17 (Estimated); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Severe Pneumonia
Keywords: pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study is a prospective observation study for lower respiratory tract infections in medical intensive care unit. Microbiologic and clinical characteristics and outcomes of patients with severe pneumonia in medical intensive care unit will be monitored and analyzed.

DETAILED DESCRIPTION:
All patients admitting medical ICU will be monitored for pneumonia. Both community-acquired (including health-care associated pneumonia) and hospital-acquired pneumonia will be included. Collecting data will include patient demographic characteristics, clinical features, microbiological characteristics including molecular work, and outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitting medical ICU with pneumonia
* Medical ICU admitted patients who is developed new pneumonia

Exclusion Criteria:

* Patients already treated more than 48 hours for pneumonia in transferring hospital and no causative organism is isolated

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitting or admitted in medical ICU with pneumonia
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2010-03; Primary Completion 2028-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Identification of etiology of pneumonia | 7 day from the time of pneumonia diagnosis

SECONDARY OUTCOMES:
Pneumonia-related death | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Ho Choi, MD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea